CLINICAL TRIAL: NCT02214745
Title: Demographic Characteristics of Children Suffering From Mental Retardation or Cerebral Palsy in the Israeli Arab Community
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0032-14-HYMC
Record Dates: First submitted 2014-08-11; First posted 2014-08-12 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Mental Retardation; Cerebral Palsy
Keywords: Israeli Arab population; Israeli/ethnology
MeSH Terms: conditions — Intellectual Disability; Cerebral Palsy | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Mentally retarded Israeli Arab children
  Interventions: Other: Questionnaire
- Israeli Arab children with cerebral palsy
  Interventions: Other: Questionnaire
- Israeli Jewish children with cerebral palsy
  Interventions: Other: Questionnaire
- Mentally retarded Israeli Jewish children
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire developed for this purpose by the investigators

SUMMARY:
To evaluate the demographic characteristics of patients suffering from mental retardation or cerebral palsy in the Israeli Arab community. Specific questionnaires will be developed and will be distributed amongst this population in order to identify these characteristics.

ELIGIBILITY:
Inclusion Criteria:

* cerebral palsy
* mental retardation
* Israeli Arab
* Israeli Jewish

Exclusion Criteria:

* all others

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Israeli Arab and Israeli Jewsih children suffering from mental retardation or cerebral palsy who have presented at the Child Development Institute at the Hillel Yaffe Medical Center.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Demographic Characteristics | One day
  Demographic characteristics will be identified through a questionnaire and will be compared with control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Mahajnah, MD, PhD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel